CLINICAL TRIAL: NCT03381690
Title: The Influence of Preoperative Epidural Labor Analgesia on Postoperative Pain in Parturients Undergoing Cesarean Section: a Retrospective Analysis
Brief Title: Preoperative Epidural Labor Analgesia and Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principle investigator, Seoul National University Bundang Hospital
Other Study IDs: Csec postop pain
Record Dates: First submitted 2017-10-24; First posted 2017-12-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epidural (ED) emergent C-sec
  Interventions: Procedure: Epidural labor analgesia
- Non-ED emergent C-sec
- Non-ED elective C-sec

INTERVENTIONS:
Procedure: Epidural labor analgesia — Epidural catheter was inserted for labor analgesia using an 18-gauge Tuohy needle and a 20 gauge epidural catheter. In our institute, for epidural labor analgesia, 10 ml bolus of 0.075% levobupivacaine mixed with fentanyl 2 μg/ml was administered and same regimen was continuously infused by patient-controlled epidural analgesia (infusion rate : 10 ml/hr, bolus : 4 ml, lockout time: 30 min).
  Groups: Epidural (ED) emergent C-sec

SUMMARY:
Parturients who undergo emergency Cesarean section (C-sec) after experiencing labor pain are likely to develop pain-induced central sensitization. The investigators hypothesized that those without epidural labor analgesia undergoing subsequent emergency C-sec would experience more severe postoperative pain or require more analgesia after C-sec compared to those with epidural labor analgesia. Thus, the investigators conducted this retrospective study by grouping parturients undergoing emergency C-sec after experiencing labor pain into two groups (epidural labor group and no epidural labor group) and those undergoing elective C-sec aimed to compare the effect of epidural labor analgesia on postoperative pain severity and analgesic consumption.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section(C-sec) under spinal anesthesia

Exclusion Criteria:

* Patients without accurate medical records
* Failure of epidural analgesia

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent elective or emergent Cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
The change of numerical rating scale for postoperative pain | At postoperative 6h, 24h, 48h, and 72h.

SECONDARY OUTCOMES:
The change of postoperative analgesic consumption | At postoperative 6h, 24h, 48h, and 72h.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea